CLINICAL TRIAL: NCT00173446
Title: Expression of D2-Like Dopamine Receptor of Human Aldosterone-Producing Adenoma and Its Role in Regulation of Aldosterone Secretion and Cell Proliferation
Brief Title: D2 Dopamine Receptor on Human Aldosterone-Producing Adenoma and Its Role in Aldosterone Secretion and Cell Proliferation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700673
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2007-06-08 (Estimated); Status verified 2005-08

CONDITIONS: Hypertension; Adrenal Aldosterone-Producing Adenoma
Keywords: Normal part of the adrenal gland
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Dopamine (DA) is one of the main catecholamines in mammals. Its major role as a brain neurotransmitter is well known as well as its contribution to the development of pathologies, mainly arterial hypertension. Traditionally, dopamine receptors are divided into two families according to the stimulation or inhibition they may produce at the adenyl cyclase level. Five dopamine receptors have been identified: D1 (D1a) and D5 (D1b) exist in the D1 family. D2s, D2l, D3 and D4 belong to the D2 family. Formerly, less than 1% of patients with hypertension were believed to have primary hyperaldosteronism; however, recent studies have suggested that primary aldosteronism affects 5-13% of patients with hypertension and aldosteronomas are a more common cause of hypertension than previously thought. At least 2% of patients with hypertension may have an aldosteronoma. The investigators' previous clinical observation found two subtypes of aldosterone-producing adenoma (APA), which were defined according to their responses to metoclopramide during salt manipulation. On a high-salt diet (HS), the nonsuppressible subjects, with less dopaminergic inhibition of aldosterone secretion, had less urinary DA excretion and greater blood pressure (BP) elevation [Wu KD et al. 2002]. The investigators' recent study of six patients with an APA found that the expression of the D2 receptor in APA was not universal. The amounts of D2 receptor messenger ribonucleic acid (mRNA) were more variant in either APA or their remnant adrenal glands. Only two cases of APA expressed the D2 receptors with much weaker signals compared with those in their respective remnant adrenals [Wu KD et al. 2001]. The investigators' current work demonstrates that the D2 receptor negatively regulates AII-stimulated aldosterone secretion and aldosterone synthase mRNA expression in NCI-H295R cells. On the other hand, the D4 receptor counteracts with the effect of the D2 receptor. In a future study, the investigators wish to quantify D2 and D4 receptor mRNA and protein expression in APA and their remnant adrenal glands and correlate them to their clinical metoclopramide test results. The investigators also wish to know whether the difference between the D2 and D4 receptor expression reflect the different effects of dopamine inhibition on AII-stimulated aldosterone secretion and aldosterone synthase transcription. Finally, the investigators will explore the role of D2 and D4 receptors on AII-stimulated adrenal cell proliferation.

ELIGIBILITY:
Inclusion Criteria:

* Adrenal aldosterone-producing adenoma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2002-01

CONTACTS AND LOCATIONS:
Overall Officials: Hong-Wei Chang, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan